CLINICAL TRIAL: NCT00939224
Title: Calibration and Validation of the a Non-Invasive Regional Oxygen Saturation Device in Neonates, Infants and Children Undergoing Cardiac Catheterization
Brief Title: Study of Non-Invasive Regional Oxygen Saturations in Pediatric Patients Undergoing Cardiac Catheterization
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP1542
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease
Keywords: Near-infrared spectroscopy (NIRS); Regional oxygen saturation; Pediatrics; Cardiac catheterization; Congenital heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort Phase 1: Cardiac Catheterization
  Interventions: Device: Model 7600 Regional Oximeter System

INTERVENTIONS:
Device: Model 7600 Regional Oximeter System — Non-invasive regional oxygen saturation measurements

SUMMARY:
The purpose of this study is to validate the Nonin Near-infrared spectroscopy (NIRS) device to measure regional oxygen saturation in a cohort of children with cardiovascular disease undergoing cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female;
* The subject is of any racial or ethnic group;
* The subject is between 0 days and 12 years of age;
* Is less than 40 kg;
* The subject is scheduled for a cardiac catheterization for treatment or diagnosis of a cardiovascular disease;
* The scheduled cardiac catheterization includes catheter placements in the central venous circulation and central arterial circulation, or catheter placement in the central venous circulation with a pre-existing arterial catheter;
* The subject is American Society Anesthesiologist (ASA) status 1 through 4; and
* The subject's legally authorized representative has given written informed consent to participate in the study and, when appropriate, the subject has given assent to participate.

Exclusion Criteria:

* Is greater than twelve (12) years of age;
* Has pre-existing allergies to adhesive tapes or adhesives on neonatal ECG pads;
* Has pre-existing skin condition at the site where the Nonin cerebral oximeter sensor will be placed (e.g., eczema, dermatitis);
* Has craniofacial disease preventing application of the sensor to the forehead;
* Has sickle cell anemia or other hemoglobinopathy;
* Has disease of the cerebrovasculature including the jugular or carotid vessels;
* Was previously on ECMO involving the carotid or jugular vessels that could have resulted in disease or ligation;
* Is not able to be in a supine position with cardiac catheterization laboratory table angle zero degrees with a neutral neck position at zero degrees rotation;
* Has acute neurological injury (seizure, stroke, encephalopathy, meningoencephalitis currently or within the past 10 days), or a structural brain lesion (eg, arteriovenous malformation, cyst) in the optical field beneath the sensor;
* Has an emergency, life-threatening condition (American Society of Anesthesiologists Physical status 5 or 6) impacting the ability to obtain informed consent;
* Or has another condition, which in the opinion of the principal investigator would not be suitable for participation in the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with cardiovascular disease (acquired or congenital; cyanotic or acyanotic; unrepaired, palliated or fully repaired) requiring cardiac catheterization to diagnose or treat the disease will be eligible for study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The success of the validation and calibration will be assessed through the Arms statistic. | Single visit

SECONDARY OUTCOMES:
Tissue (somatic) sensor readings will be described using the descriptive statistics. | Single Visit

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Mitchell, RN, BSN, Study Director — Nonin Medical, Inc
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Kreeger RN, Ramamoorthy C, Nicolson SC, Ames WA, Hirsch R, Peng LF, Glatz AC, Hill KD, Hoffman J, Tomasson J, Kurth CD. Evaluation of pediatric near-infrared cerebral oximeter for cardiac disease. Ann Thorac Surg. 2012 Nov;94(5):1527-33. doi: 10.1016/j.athoracsur.2012.05.096. Epub 2012 Aug 2. PMID 22858270